CLINICAL TRIAL: NCT05904990
Title: High-intensity Laser Therapy Improves Pain, Health Status and Quality of Life in Women With Fibromyalgia: A Single Blinded-randomized Controlled Trial
Brief Title: High-intensity Laser Therapy Improves Pain, Health Status and Quality of Life in Women With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Kerolous Ishak Shehata, principle investigator, October 6 University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: p.t.REC\012\004507
Record Dates: First submitted 2023-06-07; First posted 2023-06-15 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Intervention Model Description: High intensity laser
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- traditional exercise therapy only (Experimental): This 50-minute program included a 10-minute warm-up phase (treadmill walking at a comfortable speed), 30 minutes of stretching exercises for (glutei, paraspinal muscles, hamstring, pectoralis, scalenus, intercostal muscles, and trapezius), and a 10-minute cool-down involving self-stretching and respiratory exercises.
  Interventions: Device: traditional exercise therapy only
- HILT alongside traditional exercise therapy, (Experimental): pulsed Nd: YAG laser device (HIRO 3.0; ASA Laser, Arcugnano, Italy). This equipment delivers pulsed laser light at a wavelength of 1,064 nm, with a very high peak power of 3 kW and energy density ranging from 360 to 1,780 mJ/cm2.
  Interventions: Device: traditional exercise therapy only; Device: HILT alongside traditional exercise therapy

INTERVENTIONS:
Device: traditional exercise therapy only — 50-minute program included a 10-minute warm-up phase (treadmill walking at a comfortable speed), 30 minutes of stretching exercises for (glutei, paraspinal muscles, hamstring, pectoralis, scalenus, intercostal muscles, and trapezius), and a 10-minute cool-down involving self-stretching and respiratory exercises
Device: HILT alongside traditional exercise therapy — YAG laser device (HIRO 3.0; ASA Laser, Arcugnano, Italy). This equipment delivers pulsed laser light at a wavelength of 1,064 nm, with a very high peak power of 3 kW and energy density ranging from 360 to 1,780 mJ/cm2. It operates with short pulse durations between 120 and 150 μs, at low frequencies of 10 to 40 Hz, and has a duty cycle of about 0.1%.
  Arms: HILT alongside traditional exercise therapy,

SUMMARY:
This study will be conducted to investigate High-intensity laser therapy improves pain, health status and quality of life in women with fibromyalgia

ELIGIBILITY:
Inclusion Criteria:

1. WPI ≥ 7/19 pain sites and SSS ≥ 5/12 or WPI between > 3-6/19 and SSS > 9/12
2. symptoms have been present at a similar level for at least 3 months
3. the patient does not have another disorder that would otherwise sufficiently explain the pain
4. generalized pain, defined as pain in at least four of five regions, is present

Exclusion Criteria:

* uncontrolled diabetes
* known history of cancer

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2023-01-29 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Revised Fibromyalgia Impact Questionnaire (FIQR) | up to 6 weeks
  assesses the overall severity of FM and health status based on participant ratings. It encompasses three key domains similar to the FIQ (function, overall impact, and symptoms), with additional inquiries regarding memory, tenderness, balance, and environmental sensitivity
Visual Analog Scale (VAS) | up to 6 weeks
  10 cm, where patients rated their pain on a scale from 0 ("no pain") to 10 ("extremely severe pain ") over the past 3 days
pressure algometer | up to 6 weeks
  This tool comprises a circular rubber tip (1 cm2) and a pressure gauge for displaying readings in kilograms. Given the rubber tip's 1 cm² area, measurements were reported in kilograms per square centimeter (kg/cm2). The algometer has a measurement range from 0 to 10 kg, with increments of 0.1 kg. The instrument was pressed against the skin's surface at a right angle, and the force exerted was registered on a manometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Kerolous Ishak Shehata Kelini, Giza, Egypt